CLINICAL TRIAL: NCT07395830
Title: Effects of a Multisensory VR Experience on Stress and User Experience: A Randomized Controlled Study
Brief Title: Effects of a Multisensory VR Experience on Stress and User Experience
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Guillermo Palacios, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UTI-VI-060-2025
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: To Evaluate the Main Effects of Varying Auditory Stimuli; To Evaluate the Main Effects of Varying Olfactory Stimuli

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control Group
- Experimental (Experimental): Experimental Group
  Interventions: Other: Relaxing aroma and state of stress/calm

INTERVENTIONS:
Other: Relaxing aroma and state of stress/calm — A 2×2 randomized design is used. The Aroma condition is between subjects (relaxing aroma vs. no aroma) (experimental group and control group). The Mode condition is within each group and consists of two blocks: Stress and Calm. The order of the blocks is counterbalanced (Stress-Calm/Calm-Stress): half of the participants experience Stress first and then Calm, and the other half in the reverse order.
  Arms: Experimental

SUMMARY:
This study explicitly tests a multisensory virtual reality experience that combines visual, auditory, and olfactory channels to modulate the stress response in young adults. In addition to visual and auditory stimulation, the study also assesses whether a relaxing olfactory stimulus attenuates this effect. The environment and task remain constant (constant visuals); auditory and olfactory elements are varied. Objective. To evaluate the main effects of varying auditory and olfactory stimuli, as well as their interaction, on variables related to the performance of a quiz-type task in virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* must meet the required age.
* must have corrected vision/hearing.

Exclusion Criteria:

* uncontrolled asthma.
* uncontrolled odor-triggered migraines.
* pregnancy state.
* nasal congestion.
* severe predisposition to dizziness in virtual reality.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
NASA Task Load Index | From enrollment to the end of treatment at 2 weeks
  This test measures perceived mental workload. It has the following dimensions: Mental demand, effort, physical demand, performance, time constraints, and frustration level. Scoring interpretation:
  Higher scores for mental demand, effort, physical demand, time constraints, and frustration level indicate a greater workload/demand.
  Higher performance indicates a better experience. Reference: S. G. Hart y L. E. Staveland, "Development of NASA-TLX (Task Load Index): Results of Empirical and Theoretical Research", en Advances in Psychology, vol. 52, North-Holland, 1988, pp. 139-183. doi: 10.1016/S0166-4115(08)62386-9.
Short Stress State Questionnaire (SSSQ) | From enrollment to the end of treatment at 2 weeks
  Test to measure stress levels. It has three dimensions: engagement, anxiety, and worry. Scoring interpretation:
  * Higher score in anxiety/worry -> worse (more stress)
  * Higher score in engagement -> better (more involvement/functional activation)
  Reference: W. S. Helton y K. Näswall, "Short Stress State Questionnaire", Eur. J. Psychol. Assess., vol. 31, n.o 1, pp. 20-30, jun. 2015, doi: 10.1027/1015-5759/a000200.

SECONDARY OUTCOMES:
IPQ - Igroup Presence Questionnaire | From enrollment to the end of treatment at 2 weeks
  A test that measures overall presence in VR. Dimensions: Spatial presence, engagement, realism. Scoring logic: Higher scores indicate greater presence.
  Reference: T. Schubert, F. Friedmann, and H. Regenbrecht, "The Experience of Presence: Factor Analytic Insights," Presence Teleoperators Virtual Environ., vol. 10, no. 3, pp. 266-281, June 2001, doi: 10.1162/105474601300343603.
VRSQ - Virtual Reality Sickness Questionnaire | From enrollment to the end of treatment at 2 weeks
  It measures Cybersickness / motion sickness symptoms. Dimensions: General malaise, vestibular symptoms. Scoring logic: Higher scores indicate greater malaise.
  Reference: H. K. Kim, J. Park, Y. Choi, and M. Choe, "Virtual reality sickness questionnaire (VRSQ): Motion sickness measurement index in a virtual reality environment," Appl. Ergon., vol. 69, pp. 66-73, May 2018, doi: 10.1016/j.apergo.2017.12.016.
VAS Scale | From enrollment to the end of treatment at 2 weeks
  It measures:
  * Odor intensity (experimental only)
  * Odor liking (experimental only)
  * Odor familiarity (experimental only)
  * Perceived time pressure (both groups) Meaning: Higher scores indicate greater perceived intensity/liking/familiarity/pressure (depending on the item).
  Reference: M. Koo y S.-W. Yang, "Visual Analogue Scale", Encyclopedia, vol. 5, n.o 4, nov. 2025, doi: 10.3390/encyclopedia5040190.
UEQ-S - User Experience Questionnaire Short | From enrollment to the end of treatment at 2 weeks
  It masures the user experience. Dimensions: Pragmatic and hedonic. Scoring logic: Higher scores indicate better user experience.
  Reference: M. Schrepp, A. Hinderks, and J. Thomaschewski, "Design and Evaluation of a Short Version of the User Experience Questionnaire (UEQ-S)," Int. J. Interact. Multimed. Artif. Intell., vol. 4, no. 6, pp. 103-108, Dec. 2017.
Performance rate | From enrollment to the end of treatment at 2 weeks
  Measures of the number of correct answers, response time, and use of clues

IPD SHARING:
Plan to Share IPD: No